CLINICAL TRIAL: NCT03700788
Title: Use of 2% Chlorhexidine (CHX) as Intracanal Medicament in Endodontic Emergencies and to Compare Its Use and Effectiveness With CaOH2 (CH) Calcium Hydroxide Paste
Brief Title: 2% Chlorhexidine (CHX) vs CaOH2 (CH) Calcium Hydroxide Paste as an Intracanal Medicament
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Ramon Roges, Associate Professor, Director, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-17-00292
Record Dates: First submitted 2018-06-05; First posted 2018-10-09 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Apical Periodontitis
MeSH Terms: conditions — Periapical Periodontitis | interventions — Chlorhexidine; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant will be unaware as to which medication is used in the treatment procedure and will also be self-reporting outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clorhexidine (Experimental): 2% Chlorhexidine
  Interventions: Drug: Chlorhexidine
- Calcium Hydroxide (Active Comparator): Calcium Hydroxide
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Drug: Chlorhexidine — 2% Chorhexidine (intracranial; remains in canal until removal at next visit)
  Arms: Clorhexidine
Drug: Calcium Hydroxide — Calcium Hydroxide (intracranial; remains in canal until removal at next visit)
  Arms: Calcium Hydroxide

SUMMARY:
This is a Pilot Phase III single-blind randomized controlled clinical trial in patients, aged 18 years and older, presenting with symptoms of apical periodontitis. The overall goal is to assess whether 2% Chlorhexidine (CHX) is superior to Calcium Hydroxide in reducing interappointment pain.

DETAILED DESCRIPTION:
This is a Pilot Phase III single-blind randomized controlled clinical trial in patients, aged 18 years and older, presenting with symptoms of apical periodontitis. Patients will be treated with one of two current clinically-used medications, 2% chlorohexidine (intervention) vs. calcium hydroxide (standard-of-care). One week following treatment (+/- 2 days), patients will return for reevaltuion of apical periodontitis symptoms, via patient's pain perception after a bite test.

The primary objective of the proposed study is to determine if there is a difference in 7-day (+/- 2) post-procedure apical periodontitis following randomization to either 2% chlorohexidine vs. calcium hydroxide paste among patients presenting with symptoms of apical periodontitis. Additionally, the investigators will assess the number of adverse events that occur in each treatment group to determine if there appears to be a difference across groups, descriptively.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* symptomatic apical periodontitis (positive to the bite test)
* restorable tooth
* requires root canal therapy
* able to undergo informed consent process
* must be English or Spanish speaker

Exclusion Criteria:

* Cracked tooth
* non-restorable tooth
* no pain medication or antibiotic taken in the past 3 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
2% Chlorhexidine (CHX) vs CaOH2 (CH) Calcium Hydroxide Paste as an Intracanal Medicament. | 7 days (+/- 2 days) post treatment
  The endpoint for the proposed study will be self-reported pain post-bite test, as recorded on the visual analog scale (VAS) 7 (+/- 2) days post treatment. We will be using the Visual Analog Scale (range 1-100) and plan to analyze this as a continuous variable to maintain maximum statistical power.

SECONDARY OUTCOMES:
Is 2% Chlorhexidine (CHX) better than Calcium Hydroxide in terms of producing fewer adverse events? | 7 days (+/- 2 days) post treatment
  Secondarily, we will evaluate descriptively the proportion of adverse events in the two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Roges, D.D.S., Study Director — Director, Advanced Endodontics
Locations (1):
- Herman Ostrow USC School of Dentistry, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No